CLINICAL TRIAL: NCT05107258
Title: A Clinical Evaluation of Pine Trees Health Test System Including the Pine Trees Health Reader and COVID-19 Test for Point-of-Care
Status: Completed | Type: Observational
Sponsor: Pine Trees, Inc. (Industry)
Collaborators: Eastside Research Associates (Unknown); ICON plc (Industry); ASCLEPES Research Center (Unknown); DuPage Medical Group (Other); MRI Global (Industry); Piedmont Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: PTH-1233-01
Record Dates: First submitted 2021-11-02; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: SARS (Severe Acute Respiratory Syndrome); Covid19
Keywords: COVID-19; SARS COV-2
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Anterior nares nasal swabs in VTM.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects Symptomatic for COVID-19: Subjects must present with 1 or more of the following signs or symptoms:
  1. Fever
  2. Cough
  3. Shortness of Breath
  4. Difficulty Breathing
  5. Muscle Pain
  6. Headache
  7. Sore Throat
  8. Chills
  9. New Loss of Taste or Smell
  10. Congestion
  11. Runny Nose
  12. Diarrhea
  13. Nausea or vomiting 2. Subjects must have experienced symptom onset within the previous 10 days
  Interventions: Diagnostic Test: The Pine Trees Health Test System

INTERVENTIONS:
Diagnostic Test: The Pine Trees Health Test System — Consists of the Pine Trees Health Reader and the Pine Trees Health COVID-19 Test Kit, which contains the Pine Trees Health Cartridge, Pine Trees Health Sample Vial containing Sample Lysis Buffer and the Pine Trees Health Nasal Swab (anterior nares) for collection. The Test System is a point-of-care test used for the qualitative detection of nucleic acid from SARS-CoV-2 viral RNA in nasal swabs taken from individuals who are suspected by a healthcare professional of having COVID-19. The COVID-19 test is a rapid molecular, in vitro diagnostic test using isothermal nucleic acid amplification technology and detection of the resulting amplicon using CRISPR-mediated collateral reporter unlocking.

SUMMARY:
The scope of this study is to validate the Pine Trees Health COVID-19 Molecular Test with unique clinical specimens from across two (2) geographically diverse point-of-care testing sites in the United States. The results will be analyzed and compared against results from the CDC 2019- Novel Coronavirus (2019-nCoV) Real-Time RT-PCR Diagnostic Panel. The primary objective is to generate clinical performance data for the Pine Trees Health COVID19 molecular diagnostic test in the point-of-care setting.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is an infectious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The disease was first identified in December 2019 in Wuhan, the capital of China's Hubei province, and has since spread globally, resulting in the ongoing 2019-20 (and now 2021) coronavirus pandemic. The first confirmed case of what was then an unknown coronavirus was traced back to November 2019 in Hubei. Common symptoms include fever, dry cough, fatigue, sputum production, loss of smell, and shortness of breath. While the majority of cases result in mild symptoms, some cases progress to viral pneumonia and multi-organ failure. Emergency symptoms include difficulty breathing, persistent chest pain or pressure, confusion, difficulty waking, and bluish face or lips. The time from exposure to onset of symptoms is typically around five days but may range from two to fourteen days.

As of December 4th, 2020, more than 67.3 million cases have been reported across 185 countries and territories, resulting in more than 1.54 million deaths. On December 2nd, 2020 the Pfizer/BioNTech vaccine was approved in the United Kingdom, followed by approval in the United States (under Emergency Use Authorization [EUA]) on December 11th , 2020. Numerous antiviral and anti-inflammatory treatments have been proposed for COVID-19. Today, management involves the treatment of symptoms, supportive care, isolation, and experimental measures. The WHO has published several testing protocols for the disease [7]. The standard method of testing is real-time reverse transcription polymerase chain reaction (rRT-PCR). The test is typically done on respiratory samples obtained by a nasopharyngeal swab and more recently mid-turbinate and anterior nares nasal swab, and sputum sample or saliva may also be used. Results are generally available within 12-18 hours but can take upwards of two - four days depending on the testing needs of the community. Blood tests can be used, but these require two blood samples taken two weeks apart, and the results have little immediate value. Blood tests can be used to detect antibodies to the virus. The FDA in the United States authorized under EUA the first antigen point-of-care test on 21 March 2020 for use at the end of that month and more recently Lucira has received EUA authorization for at-home-testing.

The FDA has continued to request novel, molecular diagnostic tests which can be offered as point-of-care tests with the potential for future at-home use with a prescription. Pine Trees Health believes our Pine Trees Health Test System offers an important improvement to the global testing challenge, providing a state-of-the-art CRISPR-based test for detecting SARS-CoV-2 with sensitivity comparable to the gold standard RT-qPCR (Limit of Detection of 300 copies/mL, sensitivity >95%, specificity >99%). The Pine Trees Health Test System thus offers a low-cost and scalable alternative which will be utilized in this clinical study protocol and enable our EUA submission based on the data generated.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must present with 1 or more signs or symptoms of COVID-19 infection*.
2. Subjects must have experienced symptom onset within the previous 10 days.
3. Subject or Subject's legally authorized representative (LAR) is willing and able to provide informed consent. Adult subjects unable to consent will provide assent in addition to LAR's consent.
4. Subject is ≥ 6 years of age. Subjects 6 ≥ x ≤ 17 will provide assent in addition to parent/legal guardian's consent.

Exclusion Criteria:

1. Individual is not able to tolerate sample collection.
2. The subject has been positive for SARS-CoV-2 previously.
3. The subject underwent a nasal wash/aspirate as part of standard of care <24 hours prior to the study visit.
4. The subject is currently receiving or has received within the past thirty (30) days of the study visit an experimental biologic, drug, or device including either treatment or therapy.
5. The subject has previously participated in this research study.

   * Symptoms may appear 2-10 days after exposure and may include one or more of the following: Fever, Cough, Shortness of Breath, Difficulty Breathing, Muscle Pain, Headache, Sore Throat, Chills, New Loss of Taste or Smell, Congestion, Runny Nose, Diarrhea, Nausea or vomiting.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals symptomatic of COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | Two weeks
  The primary outcome of our study will be to determine the positive and negative comparator agreement (PPA and NPA), sensitivity and specificity of the Pine Trees Health COVID-19 diagnostic test.

SECONDARY OUTCOMES:
Secondary Outcome | Two Weeks
  The secondary objective of this study is to determine the likelihood ratio of positive predictive value to likelihood ratio negative predictive value, standard positive predictive value and standard negative predictive value.

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Milos, PhD, Study Director — Pine Trees Health
Locations (3):
- United States (3):
  - ASCLEPES Research Center, Spring Hill, Florida
  - PMG Research of Piedmont Healthcare, Statesville, North Carolina
  - Eastside Research Associates, Redmond, Washington

IPD SHARING:
Plan to Share IPD: No
No plan, subjects will be de-identified and data will only be going to the sponsor.